CLINICAL TRIAL: NCT06947187
Title: Vaccine Confidence and Infodemic in Southeast Asia's Nusantara Sociocultural Sphere: A Transdisciplinary, Transnational Study
Brief Title: Vaccine Confidence and Infodemic in Southeast Asia's Nusantara Sociocultural Sphere
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Laura (Layla) H Kwong, Assistant Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-06-16452
Record Dates: First submitted 2025-01-06; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Misinformation
Keywords: Misinformation; Bahasa; Vaccine confidence; Vaccine literacy; Video intervention
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watch pre-bunking video (Experimental): Participants in this arm will watch a ~3-minute pre-bunking video
  Interventions: Other: Pre-bunking video
- Watch video on safe disposal of medication (Placebo Comparator): Participants in this arm will watch a ~3-minute video that discusses safe ways to dispose of medication
  Interventions: Other: Video on safe disposal of medication

INTERVENTIONS:
Other: Pre-bunking video — ~3 minutes educational video to improve vaccine literacy and vaccine confidence
  Arms: Watch pre-bunking video
Other: Video on safe disposal of medication — ~3 minutes educational video on safe disposal of medication
  Arms: Watch video on safe disposal of medication

SUMMARY:
The goal of this clinical trial is to understand how well a culturally-specific "prebunking" video can improve vaccine information literacy and vaccine confidence among individuals in the Nusantara sociocultural sphere. The investigators hypothesize the individuals who watch the co-created "prebunking" intervention video will have improved vaccine literacy skills and vaccine confidence compared to individuals who watch a video about safe medication disposal.

DETAILED DESCRIPTION:
The primary aim of this research is to develop and assess the impact of an educational video in enhancing vaccine information literacy and vaccine confidence within Southeast Asia's Nusantara Sociocultural Sphere--a network of communities spanning multiple countries in Southeast Asia, connected by shared linguistic, historical, and sociocultural roots. Adopting a transdisciplinary and human-centered approach, we will engage representatives from Brunei, Indonesia, Malaysia and Singapore through online workshops and in-person focus group discussions to co-create a video. Guided by the findings from our research (using publicly available social media dataset) and communication theories from existing literature, the video will contain messages that focus on equipping viewers with the skills to identify common tactics used in vaccine misinformation in two mutually intelligible languages (Bahasa Melayu and Bahasa Indonesia) and on enhancing vaccine confidence levels among viewers.

To evaluate the effectiveness of the videos as an intervention for vaccine information literacy and vaccine confidence, we will conduct an online two-arm randomized controlled trial (RCT). Participants will be randomly assigned to one of the two groups:

1. Group 1 (Intervention Group): Participants will watch the co-created video containing vaccine-related messages.
2. Group 2 (Control Group): Participants will watch a control video containing messages related to the importance of proper and safe medication disposal.

We hypothesize that exposure to Video 1 will lead to a significant increase in vaccine literacy skills and vaccine confidence compared to exposure to Video 2.

The study will be conducted online. Individuals who have signed the e-consent form will be automatically redirected to the online RCT. Each participant will be asked to respond to several pre-video questions (including demographic, vaccine confidence, and vaccine literacy). After stratification by language, they will be randomly assigned to watch either the control video (physical exercise) or intervention video (vaccine) using REDCap's randomization functionality. After watching the video, they will respond to post-video questions (including behavior, vaccine confidence, and vaccine literacy). They will then undergo debriefing, which aims to clarify which social media posts (embedded in vaccine literacy-related questions) contain misinformation AND to provide full disclosure on the goal of the RCT (which was partially disclosed during recruitment to avoid confusion). Finally, each participant will be asked if they are interested to participate in a gift card drawing -- if they are, the investigators will asked them to share their name and contact information. The UCB team will monitor data collection and stop data collection when the target number of participants has been reached.

Within two weeks of closing the RCT data collection, the UCB team will draw 40 names from a pool of participants who have successfully completed the experiment and have agreed to participate in the drawing for gift cards. 20 out of 40 selected participants will be from the Bahasa Melayu-speaking pool; the other 20 from the Bahasa Indonesia-speaking pool.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Live in Brunei, Indonesia, Malaysia, or Singapore
* Fluent in Bahasa Melayu or Bahasa Indonesia
* Watch social media content in Bahasa Melayu or Bahasa Indonesia every day
* Access to stable Internet on smartphone or laptop to complete the experiment without interruption

Exclusion Criteria:

* Individuals who were involved in the online human-centered design thinking workshops or the in-person focus-group discussions will not be eligible to participate in RCT. This exclusion criterion is put in place to prevent potential bias in the evaluation of the intervention's effectiveness.
* Individuals who have difficulty in looking at social media on cellphone (even when they use prescription glasses), listening to the audio of social media content on cellphone (even with hearing aid), and typing within or engaging with social media content on cell phone are not eligible to participate in this study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of vaccine misinformation | From the start to the end of the survey (approximately 20 minutes)
  The percent of social media posts that the participant correctly identifies as misinformation

SECONDARY OUTCOMES:
Vaccine confidence | From the start to the end of the survey (approximately 20 minutes)
  The participant's stated vaccine confidence on a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Laura H Kwong, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No